CLINICAL TRIAL: NCT01033084
Title: A Factorial, Double-blinded, Randomized Clinical Trial on Major Depressive Disorder Using Transcranial Direct Current Stimulation
Brief Title: Efficacy Study of Transcranial Direct Current Stimulation to Treat Major Depressive Disorder
Acronym: SELECT-TDCS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Andre Brunoni, MD, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USP-HU-001; FAPESP2009/05728-7 (Other Grant/Funding Number: FAPESP 2009/05728-7)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sham stimulation / sertraline (Experimental): In this arm, patients will receive sham stimulation and sertraline 50mg/day. In sham stimulation, the tDCS device is set in the same fashion as the active stimulation, but the device is turned off after one minute of stimulation.
  Interventions: Drug: Sertraline
- Sham stimulation / placebo pill (Sham Comparator): Placebo pills are sugar pills having the same size and shape of the active pills.
  In sham stimulation, the tDCS device is set in the same fashion as the active stimulation, but the device is turned off after one minute of stimulation.
  Interventions: Other: double placebo
- Active stimulation / Sertraline (Experimental): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp (which is located on the intersection of the sagittal and median curves). The device will deliver a charge of 2mA for 30 minutes.
  Patients will receive Sertraline 50mg/day.
  Interventions: Device: transcranial direct current stimulation; Drug: Sertraline
- Active stimulation / placebo pill (Experimental): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp (which is located on the intersection of the sagittal and median curves). The device will deliver a charge of 2mA for 30 minutes.
  Placebo pills are sugar pills having the same size and shape of the active pill
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation will be applied at 2mA, 30 minutes/day, for 10 weekdays consecutively and two extra stimulations at week 4 and 6.
  Arms: Active stimulation / Sertraline; Active stimulation / placebo pill
Drug: Sertraline — Patient will receive sertraline 50mg/day.
  Arms: Active stimulation / Sertraline; Sham stimulation / sertraline
Other: double placebo — double placebo arm (sham stimulation/placebo pill)
  Arms: Sham stimulation / placebo pill

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation is an effective treatment for major depression, when compared (and combined) to sertraline and placebo.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a common mental disorder, with a lifetime prevalence of 15% and an incidence of 5% per year. Its core symptoms include lack of pleasure in daily activities, thoughts of guilt and depressed mood. According to the World Health Organization, MDD is one of the ten most impairing conditions, leading to missing workdays, loss of quality of life and increasing expenses in health care. Besides, about 1% of patients with MDD complete suicide. Moreover, one third of patients with MDD remain depressed after more than two adequate treatments, i.e., they are refractory to conventional antidepressant treatments; also, most treated patients remain with residual symptoms. Therefore, the development of new treatments is necessary. Transcranial direct current stimulation (tDCS) is a novel, promising technique in the study of several neuropsychiatric conditions.

Transcranial DCS is a non-invasive brain stimulation method in which a low intensity direct current is applied through the skull, with neurophysiologic studies showing that a considerable amount of electrical current reach the brain tissues, vis-à-vis the specified parameters. Thus, the DC could be applied over brain MDD-related areas, such as the dorsolateral prefrontal cortex, thereby leading to neuroplasticity and MDD treatment. Indeed, some pilot studies showed that tDCS might ameliorate depressive symptoms. However, it is necessary to replicate these findings in larger populations to increase the generalizability of the results and to verify the efficacy of the intervention. Our aim is to perform a double blind, randomized, factorial study comparing tDCS and sertraline for MDD treatment, enrolling 120 eligible patients of both genders between 21-65 years not presenting active suicidal ideation. They will be allocated in 4 groups at random to receive active tDCS or sham and sertraline 50mg/day or placebo. Transcranial DCS will be applied in a daily basis for 10 consecutive working days (2 weeks), after that, the patients will be followed weekly for 6 weeks. Our primary outcome is the depression rating scores at 6 weeks, measured by the Hamilton Depression Rating Scale (HDRS), 17-itens. In conclusion, our purpose is to perform a clinical tDCS study to verify its efficacy in the treatment of MDD in a sample of patients of several levels of severity and refractoriness.

Our secondary objectives are also to verify the safety of the intervention as well as to compare tDCMajor Depressive Disorder (MDD) is a common mental disorder, with a lifetime prevalence of 15% and an incidence of 5% per year. Its core symptoms include lack of pleasure in daily activities, thoughts of guilt and depressed mood. According to the World Health Organization, MDD is one of the ten most impairing conditions, leading to missing workdays, loss of quality of life and increasing expenses in health care. Besides, about 1% of patients with MDD complete suicide. Moreover, one third of patients with MDD remain depressed after more than two adequate treatments, i.e., they are refractory to conventional antidepressant treatments; also, most treated patients remain with residual symptoms. Therefore, the development of new treatments is necessary. Transcranial direct current stimulation (tDCS) is a novel, promising technique in the study of several neuropsychiatric conditions.

Transcranial DCS is a non-invasive brain stimulation method in which a low intensity direct current is applied through the skull, with neurophysiologic studies showing that a considerable amount of electrical current reach the brain tissues, vis-à-vis the specified parameters. Thus, the DC could be applied over brain MDD-related areas, such as the dorsolateral prefrontal cortex, thereby leading to neuroplasticity and MDD treatment. Indeed, some pilot studies showed that tDCS might ameliorate depressive symptoms. However, it is necessary to replicate these findings in larger populations to increase the generalizability of the results and to verify the efficacy of the intervention. Our aim is to perform a double blind, randomized, factorial study comparing tDCS and sertraline for MDD treatment, enrolling 120 eligible patients of both genders between 21-65 years not presenting active suicidal ideation. They will be allocated in 4 groups at random to receive active tDCS or sham and sertraline 50mg/day or placebo. Transcranial DCS will be applied in a daily basis for 10 consecutive working days (2 weeks), after that, the patients will be followed weekly for 6 weeks. Our primary outcome is the depression rating scores at 6 weeks, measured by the Hamilton Depression Rating Scale (HDRS), 17-itens. In conclusion, our purpose is to perform a clinical tDCS study to verify its efficacy in the treatment of MDD in a sample of patients of several levels of severity and refractoriness.

Our secondary objectives are also to verify the safety of the intervention as well as to compare tDCS vs. sertraline and the association of sertraline and tDCS vs. each treatment alone in major depression treatment.

ELIGIBILITY:
Inclusion Criteria:

* Depressive Disorder, Major (SCID)
* HDRS > 18

Exclusion Criteria:

* Other axis I disorders, including Bipolar Disorder, Schizophrenia, Substance Abuse Disorders.
* Any axis II disorders.
* Any serious/life-threatening axis III disorders, such as Congestive Heart Failure, Pulmonary Obstructive Chronic Disease, Active Neoplasia.
* Neurological diseases such as Stroke (and Post-Stroke Depression), Dementias and others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
MADRS score | repeated-measures

SECONDARY OUTCOMES:
HDRS-17 score at week 6. | week 6
Remission rate (MADRS<=10) | week 6
MADRS score | week 2

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Vieira GP, Bueno VF, Goulart AC, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. Sertraline vs. ELectrical Current Therapy for Treating Depression Clinical Trial--SELECT TDCS: design, rationale and objectives. Contemp Clin Trials. 2011 Jan;32(1):90-8. doi: 10.1016/j.cct.2010.09.007. Epub 2010 Sep 18. PMID 20854930
- [Background] Alessandra Baccaro, Andre Russowsky Brunoni, Isabela Martins Bensenor, Felipe Fregni. Hypomanic episode in unipolar depression during transcranial direct current stimulation. Acta Neuropsychiatrica 22(6):316-318, 2010.
- [Derived] Brunoni AR, Kemp AH, Dantas EM, Goulart AC, Nunes MA, Boggio PS, Mill JG, Lotufo PA, Fregni F, Bensenor IM. Heart rate variability is a trait marker of major depressive disorder: evidence from the sertraline vs. electric current therapy to treat depression clinical study. Int J Neuropsychopharmacol. 2013 Oct;16(9):1937-49. doi: 10.1017/S1461145713000497. Epub 2013 Jun 12. PMID 23759172
- [Derived] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Goulart A, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. The sertraline vs. electrical current therapy for treating depression clinical study: results from a factorial, randomized, controlled trial. JAMA Psychiatry. 2013 Apr;70(4):383-91. doi: 10.1001/2013.jamapsychiatry.32. PMID 23389323